CLINICAL TRIAL: NCT03345147
Title: LOAEL/NOAEL and UL Determination in Guatemala - Estimation of Vitamin A Stores in Children and Women and Correlation With Potential Toxicity Markers
Brief Title: Estimation of Vitamin A Stores in Children and Women in Guatemala and Relation With Potential Toxicity Markers
Acronym: GloVitAS-GU
Status: Completed | Type: Observational
Sponsor: Institute of Nutrition of Central America and Panama (Other)
Collaborators: Newcastle University (Other); Bill and Melinda Gates Foundation (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Dora Ines Mazariegos, MSc, Researcher, Nutritional Biochemistry Laboratory, Institute of Nutrition of Central America and Panama
Other Study IDs: CIE-REV 061/2016
Record Dates: First submitted 2017-08-25; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Vitamin A Status
Keywords: Vitamin A; Isotopic dilution; dietary assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood will be drawn on Day 4 post C-13 Vitamin A administration (women and children) and one variable day (children only) to obtain plasma, serum, and buffy coat (Day 4), or only plasma on variable day post Vitamin A dose for children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Vitamin A intake: Normal Vitamin A intake will be assessed by a questionnaire directed to the consumption of food items with high VA content on the 7 days prior to the questionnaire. The daily consumption will be assessed on average. A child is assigned to Normal Vit. A consumption if daily Vit. A is between 250 and 600 micrograms per day.
  Interventions: Other: Normal Vitamin A intake
- High Vitamin A intake: High Vitamin A intake will be assessed by a questionnaire directed to the consumption of food items with high VA content on the 7 days prior to the questionnaire. The daily consumption will be assessed on average. A child is assigned to High Vit. A consumption if daily Vit. A is above 900 micrograms per day.
  Interventions: Other: High Vitamin A intake

INTERVENTIONS:
Other: High Vitamin A intake — Total Vitamin A stores will be assessed by isotopic measurement, 13C-Retinol will be given to the subject and blood wil be drawn on Day 4 to assess the isotopic dilution in the plasma. Other biochemical indicators will be assessed too, along with Dietary assessment (Food Frequency, 24 hours recalls).
  Groups: High Vitamin A intake
Other: Normal Vitamin A intake — Total Vitamin A stores will be assessed by isotopic measurement, 13C-Retinol will be given to the subject and blood wil be drawn on Day 4 to assess the isotopic dilution in the plasma. Other biochemical indicators will be assessed too, along with Dietary assessment (Food Frequency, 24 hours recalls).
  Groups: Normal Vitamin A intake

SUMMARY:
The goal of this study is to assess whether 3-5 years-old children who have Vitamin A intakes above the tolerable upper intake level (UL=900 ug per day) have higher total body Vitamin A stores and biomarkers of excessive vitamin A status, compared to children with Normal Vitamin A intakes (250-600 ug per day).

DETAILED DESCRIPTION:
The goal of this study is to assess whether VA intakes above the tolerable upper intake level (UL) and exposure to multiple programs are associated with are associated with 1) exposure to multiple VA intervention programs, and 2) elevated liver vitamin A concentration and biomarkers of excess vitamin A. Guatemala was selected as a study site because the country has a long standing national fortification program for vitamin A in sugar (law since 1975, re-launched and maintained since the 90´s). Typically, fortified sugar is used in more than 90% of households at average concentrations of 9 to 10 µg/g of sugar. VA fortified foods, in the form of fortified sugar, foods prepared with fortified sugar and other fortified foods, reach children from 2 years old to adulthood. On the other hand, high dose VA supplements, provided by local health services, only reached 10.5% of children ages 6-59 month in 2013. Children ages 2-3 and 4-5 years old with VA intakes above and below the UL will be recruited together with their mothers to assess the cumulative effect of fortification on young children and their mothers. Data from Program of Food and Nutrition Security (PROSAN), of the Ministry of Health, Guatemala in 2013, shows that coverage in the 30 Health Areas of the country is 17.9%, the lowest is 4.4% (San Marcos) and the largest 33% (Petén). Four of the 30 Region Areas correspond to the Department of Guatemala, in which urban and peri-urban areas of Guatemala City are included. In Central and North-West Guatemala Areas, coverage is 23 and 22% respectively, both above national average coverage and within the 10 out of 30 top coverages. According to PROSAN data for Micronutrient Powders in 2013, all four regions North-East, North-West, South, and Central Guatemala areas are also around or above the national coverage (14%) with 21.8, 11.2, 17.3 and 13.8% coverage. Another advantage of remaining in the 4 areas of Health around Guatemala city is that the four combined amount for 300,000 children of 0-59 month-old, that is more than 15% of the national children population reported. Even if coverages are low, population density will easier children recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-5 years old and their mothers
* Child VA intake must be above 250 micrograms/day
* Children must be apparently healthy, Hemoglobin>9 g/dL at recruitment point, C-reactive protein<5 mg/L. For Women, Hemoglobin>10 g/dL, C-reactive protein<5 mg/L

Exclusion Criteria:

°Children with Congenital or chronical diseases, reported illnesses 1 week before the test. For Women: Pregnancy or lactation, Previously known Chronic Diseases

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and Women from Guatemala peri-urban areas or areas where High Vitamin A foods intake is reported. Convenience sampling according to the availability (time to participate in the study) of the participant, and acceptance of Blood sampling and Dietary assessments
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Total Vitamin A stores among 3-5 years-old children, in micromoles | 28-day study period
  Estimated using Carbon 13 (13C) 13C-retinol dilution method, by the ratio of Labelled (stable isotope) versus no labelled Vitamin A in plasma 4 days after dose of labelled VA is given.
Total dietary vitamin A intake among 3-5 years-old children, in micrograms (ug) | 28-day study period
  Estimated using 24-hour dietary recalls, observed weigh food records, food and supplement frequency questionnaire

SECONDARY OUTCOMES:
Plasma retinol among 3-5 years-old children | 28-day study period
  Estimated by High Performance Liquid Chromatography (HPLC)
Plasma retinol binding protein among 3-5 years-old children | 28-day study period
  Estimated by ELISA
Plasma Transthyretin among 3-5 years-old children | 28-day study period
  Estimated by immunometric automated assay
Bone Health markers among 3-5 years-old children | 28-day study period
  Estimated by different techniques
Liver function markers among 3-5 years-old children | 28-day study period
  Estimated by different techniques
Plasma retinol among women | 28-day study period
  Estimated by HPLC
Plasma retinol binding protein among women | 28-day study period
  Estimated by ELISA
Plasma Transthyretin among women | 28-day study period
  Estimated by immunometric automated assay
Total dietary vitamin A intake among women, in micrograms (ug) | 28-day study period
  Estimated using 24-hour dietary recalls, observed weigh food records, food and supplement frequency questionnaire

OTHER OUTCOMES:
Hemoglobin concentration in children | At recruitment
  Measured with Quik Read Pro portable Device
Children weight and length | At recruitment
  Measured with Scale and Measurement Rod
Systemic inflammation in children | At recruitment
  Measured with Quik Read Pro portable Device
Iron status in children | 28-day study period
  Estimated by different techniques
Zinc status in children | 28-day study period
  Estimated by atomic emission spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Dora I Mazariegos, MsSc, Principal Investigator — Institute of Nutrition of Central America and Panama
Locations (3):
- Guatemala (3):
  - Mixco, La Comunidad City Hall, Guatemala City
  - Sacatepequez City Hall, Guatemala City
  - Santa Catarina Pinula City Hall, Guatemala City

IPD SHARING:
Plan to Share IPD: Yes
All Collected individual participant data (IPD) will be shared within the researchers group of the Global Project (GLOVITAS, leaded by Newcastle University). Only initials will identify individual participants and the information shared will be on biochemical markers, diet, and general socioeconomic data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available when, after study data collection is finished, data are cleaned and analyzed.
Access Criteria: All pre-defined researchers will have access to database. This includes Georg Lietz, principal coordinator, and local Principal researchers.
URL: https://researchtools.ncl.ac.uk

REFERENCES:
- [Derived] Ford JL, Green JB, Haskell MJ, Ahmad SM, Mazariegos Cordero DI, Oxley A, Engle-Stone R, Lietz G, Green MH. Use of Model-Based Compartmental Analysis and a Super-Child Design to Study Whole-Body Retinol Kinetics and Vitamin A Total Body Stores in Children from 3 Lower-Income Countries. J Nutr. 2020 Feb 1;150(2):411-418. doi: 10.1093/jn/nxz225. PMID 31535129